CLINICAL TRIAL: NCT02636192
Title: Incidence of Diabetic Ketoacidosis Among Patients With Type 2 Diabetes Mellitus Treated With SGLT2 Inhibitors or Other Antihyperglycemic Agents- A Retrospective, Observational, New-User Cohort Study Using 4 Administrative Claims Databases in the US
Brief Title: Study on Incidence of Diabetic Ketoacidosis Among Participants With Type 2 Diabetes Mellitus Treated With Sodium-glucose Co-transporter 2 (SGLT2) Inhibitors or Other Antihyperglycemic Agents
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108054; RRA-15322 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Sodium-glucose co-transporter 2 inhibitors; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Cohort 1: Cohort 1 included participants who were exposed to sodium-glucose co-transporter 2 (SGLT2) inhibitor (canagliflozin, dapagliflozin and empagliflozin).
  Interventions: Drug: No Intervention
- Cohort 2: Cohort 2 included participants who were exposed to other non-SGLT2 antihyperglycemic agents (AHA).
  Interventions: Drug: No Intervention

INTERVENTIONS:
Drug: No Intervention — This is an observational study and participants did not receive any intervention in this study.

SUMMARY:
The purpose of this study is to compare the incidence of diabetic ketoacidosis (DKA) among participants diagnosed with type 2 diabetes mellitus (T2DM) and pair-matched on exposure propensity scores for new use of any sodium-glucose co-transporter 2 inhibitors (SGLT2i) versus new use of various other antihyperglycemic agents (AHAs), combined as one group.

DETAILED DESCRIPTION:
This study will be an overall retrospective, observational, new-user cohort study using 4 large administrative claims databases in the US. Participants diagnosed with T2DM and initiated on SGLT2i or other AHAs (metformin, sulfonylureas (SU), thiazolidinediones (TZDs), DPP-4 inhibitors (DPP4i), GLP-1 agonists, insulin, and other AHAs) between April 1, 2013 and the end of claims data availability will be included in the study and will be estimated for incidence rates of DKA in the different AHA new-user groups.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 antihyperglycemic agents (AHA) prescription (Rx) during the study period, between 4/1/2013 and 9/30/2014.
* Diagnosed of type 2 diabetes mellitus
* Enrollment history of at least 12 months
* Having prescription drug coverage
* Having no prescription of the index drug during the 6 months prior

Exclusion Criteria:

- Participants who receive diagnosis of type1 diabetes mellitus (T1DM) and/or secondary diabetes mellitus (SDM) any time after index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with type 2 diabetes mellitus (T2DM) and initiated on sodium-glucose co-transporter 2 inhibitors (SGLT2i) or other Antihyperglycemic Agents (AHAs) were observed.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with a recorded diagnosis of Diabetic Ketoacidosis (DKA) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trials, Study Director — Janssen Research & Development, LLC